CLINICAL TRIAL: NCT05244902
Title: Gastric Emptying Times of Normal and Obese Children After Preoperative Clear Fluid Drinking: An Ultrasound Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, muhammet korkusuz, Principle investigator, MD, Karaman Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-2021/12
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Gastric Emptying Time
Keywords: Gastric volume; Gastric emptying time; Antral cross-sectional area (ACSA); Obese pediatric patients
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Pediatric patients will be divided into two groups as obese and non-obese. Children above the 95% percentile will be considered as obese.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese pediatric patient (Experimental): Obese children aged 6-14 years, over 95% percentile, fasted for the night before planned surgery.
  Interventions: Drug: 5% Dextrose
- Non-obese pediatric patient (Active Comparator): Non-obese children aged 6-14 years, between 5-85% percentile, fasted for the night before planned surgery.
  Interventions: Drug: 5% Dextrose

INTERVENTIONS:
Drug: 5% Dextrose — All the patients will receive oral 3mL/kg 5%Dextrose

SUMMARY:
In the recent literature, pre-operative fasting times for pediatric patients are limited to one hour for clear fluids. Studies related to gastric emptying times mostly searched for normal-weight children. These studies have claimed that 3 mL/kg clear fluid can be allowed up to 1 hour before surgery. There is a lack of interest in the gastric emptying time of obese pediatric patients during the preoperative period. In addition, there is controversy about gastric emptying times of obese healthy children. Some research committed the decrease of gastric emptying because of a high level of sensitivity to cholecystokinin, while others postulated that no change in gastric emptying time of obese children compared to normal weight. The aim of this trial is to compare the gastric volume and gastric emptying time after ingestion of 3 mL/kg clear fluid in obese and non-obese pediatric patients in the pre-operative period.

DETAILED DESCRIPTION:
After receiving informed consent from the children and their families, American Society of Anesthesiologists (ASA) 1-2 pediatric patients between 6-14 years, who will recruit for elective surgery will be included for this study. The children over 95% percentile will be accepted as obese. After, the basal gastric volume will be calculated with the help of Ultrasonography (USG). The children will receive oral 3 mL/kg(max 250 mL) 5% dextrose .USG evaluation will be made every 5 minutes until the gastric volume reaches the basal level. Children reaching basal gastric volume will be accepted as suitable for the surgery. The aim of this study is to compare the gastric volume and gastric emptying time after ingestion of 3 mL/kg clear fluid in obese and non-obese pediatric patients in the pre-operative period.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical state I or II
* Age 6 to 14 years.
* Gender: both sexes.
* Scheduled for non-Gastrointestinal Tract elective day-case surgery under general anesthesia.

Exclusion Criteria:

* Parent/ care giver refusal
* Ages < 6 or > 14 years old
* Children with gastro-esophageal reflux disease
* Renal failure
* Diabetes mellitus
* Cerebral palsy patients
* Mental retardation
* Esophageal strictures, achalasia or any intestinal disease that may impair the gastric emptying.
* Gastrointestinal system surgery and neurosurgical patients
* Emergency surgery
* Violation of the prescribed fasting times
* Refusing to drink prescribed clear fluid

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time | 90 minute
  Time until the gastric volume reaches the baseline level again.

SECONDARY OUTCOMES:
Antral cross-sectional area | 90 minute
  Antral cross-Section Area (ACSA) (cm2) maximal anteroposterior diameter (D1) and longitudinal diameter (D2) will be measured with ultrasound and calculated with that mathematical formula:
  ACSA(cm2) = Π x D1 x D2 / 4

OTHER OUTCOMES:
Gastric emptying half-time ( t 1/2) | 90 minute
  Time required for ACSA to return to half maximum value.
Gastric volume | 90 minute
  The mathematical model will be used which was reported by Perlas and colleagues based on gastroscopic fluid assessment will be used for the calculation of gastric volume (mL) from ACSA. GastricVolume(mL) = 27.0 + 14.6 x ACSA(cm2) -1.28 x Age(years)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet Korkusuz, MD, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Taining and Research Hospital, Karaman, Turkey (Türkiye)